CLINICAL TRIAL: NCT06117826
Title: Incidince of Acute Kidney Injury in Children With Community Acquired Pneumonia at Assiut University Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ‪Mohamed Mahmoud Fathy Ahmed, 71515,Assiut, Assiut University
Other Study IDs: Incidence of kidney injury
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive prospective observational study of Incidince of acute kidney injury in children with community acquired pneumonia at assiut university children hospital

DETAILED DESCRIPTION:
Community acquired pneumonia (CAP) is a prevalent cause of infectious mortality worldwide [1, 2]. The number of patients hospitalized with CAP in the United States has been estimated to have reached one million in 2020, with similarly significant increases globally [3]. In Egypt, it was estimated that 10% of children deaths below the age of 5 years is likely caused by pneumonia and other acute respiratory infections [4] Acute kidney injury (AKI) is an abrupt decrease in glomerular filtration rate that can lead to health consequences for children in both the short and long term [5]. In fact, AKI may increase hospitalization length and morbidity and mortality rates for patients in the short term. Meanwhile, it exposes them to an increased risk of chronic kidney disease (CKD) over time. Even mild AKI doubles the risk of CKD during follow-up [6] . AKI is a common condition among hospitalized children. Reports indicate that AKI can exacerbate several typical pediatric disorders, such as acute gastroenteritis with an AKI prevalence of around 25% [7], type 1 diabetes mellitus onset with a prevalence rate of approximately 45% [8], and acute appendicitis at roughly 7% incidence levels[9] . Acute kidney injury (AKI) frequently complicates CAP; its incidence ranges from18-34 %in CAP patients[10-12]. Chawla et al., previously reported that coexisting pneumonia and AKI led to worse outcomes than either pneumonia or AKI alone[13]. Even among non-severe cases diagnosed only as pneumonia, however,Aki was associated with long-term mortality[11]. Despite this evidence, the impactof Aki on inhospital outcomes remains unclear for Egyptian populations . Adults suffering from CAP present considerable risks when it comes to developing both acute kidney injury(AKI)[14-15]and later chronic kidney disease(CKD)[16]; we hypothesize that there might be under-recognition regarding the prevalence of AKIs among children hospitalized due to CAP-especially milder forms. Indeed even milder forms double CKD risks during follow-ups.[17]Thus,it becomes crucially important to detect any episodes of Aki in order plan appropriate patient follow-ups.

ELIGIBILITY:
Inclusion Criteria:

- Patients age <18 years who are diagnosed with x-ray confirmed communityacquired pneumonia(CAP)

Exclusion Criteria:

* We excluded patients with preexistent comorbidities potentially affecting the Severity of pneumonia

Ages: 30 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children hospitalized with community-acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidince of acute kidney injury in children with community acquired pneumonia at assiut university children hospital | Baseline
  Incidince of acute kidney injury in children with community acquired pneumonia at assiut university children hospital

REFERENCES:
- [Background] GBD 2016 Causes of Death Collaborators. Global, regional, and national age-sex specific mortality for 264 causes of death, 1980-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1151-1210. doi: 10.1016/S0140-6736(17)32152-9. PMID 28919116
- [Background] Jain S, Williams DJ, Arnold SR, Ampofo K, Bramley AM, Reed C, Stockmann C, Anderson EJ, Grijalva CG, Self WH, Zhu Y, Patel A, Hymas W, Chappell JD, Kaufman RA, Kan JH, Dansie D, Lenny N, Hillyard DR, Haynes LM, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, Wunderink RG, Edwards KM, Pavia AT, McCullers JA, Finelli L; CDC EPIC Study Team. Community-acquired pneumonia requiring hospitalization among U.S. children. N Engl J Med. 2015 Feb 26;372(9):835-45. doi: 10.1056/NEJMoa1405870. PMID 25714161
- [Background] Coca SG, Singanamala S, Parikh CR. Chronic kidney disease after acute kidney injury: a systematic review and meta-analysis. Kidney Int. 2012 Mar;81(5):442-8. doi: 10.1038/ki.2011.379. Epub 2011 Nov 23. PMID 22113526
- [Background] Chawla LS, Amdur RL, Faselis C, Li P, Kimmel PL, Palant CE. Impact of Acute Kidney Injury in Patients Hospitalized With Pneumonia. Crit Care Med. 2017 Apr;45(4):600-606. doi: 10.1097/CCM.0000000000002245. PMID 28291091